CLINICAL TRIAL: NCT01004289
Title: POSTconditioning During Coronary Angioplasty in Acute Myocardial Infarction Study (POST-AMI)
Brief Title: POSTconditioning During Coronary Angioplasty in Acute Myocardial Infarction Study
Acronym: POST-AMI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Padova (Other)
Responsible Party: Giuseppe Tarantini, Department of Cardiac, Thoracic and Vascular Sciences. University of Padua
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1328P
Record Dates: First submitted 2009-10-28; First posted 2009-10-29 (Estimated); Last update posted 2010-10-15 (Estimated); Status verified 2010-10

CONDITIONS: Myocardial Reperfusion Injury
Keywords: Acute myocardial infarction; Primary percutaneous coronary intervention; Postconditioning
MeSH Terms: conditions — Myocardial Reperfusion Injury | interventions — Ischemic Postconditioning; Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator): Primary angioplasty and stenting without additional intervention.
  Interventions: Procedure: Primary angioplasty and stenting without additional intervention
- Postconditioning (Experimental): Primary angioplasty and stenting followed by brief episodes of ischemia-reperfusion performed during the first minutes of reperfusion.
  Interventions: Procedure: Postconditioning

INTERVENTIONS:
Procedure: Postconditioning — Primary angioplasty and stenting followed by brief episodes of ischemia-reperfusion performed during the first minutes of reperfusion
  Other Names: Staccato Reperfusion
  Arms: Postconditioning
Procedure: Primary angioplasty and stenting without additional intervention — Primary angioplasty and stenting without additional intervention.
  Arms: Control

SUMMARY:
The POST-conditioning during coronary angioplasty in Acute Myocardial Infarction (POST-AMI) trial will evaluate the usefulness of postconditioning in limiting infarct size and microvascular damage during the early and late phases after AMI.

DETAILED DESCRIPTION:
POST-AMI is a single-center, prospective, randomized trial, with a planned inclusion of 78 patients with ST-elevation Acute Myocardial Infarction (AMI). Patients will be randomly assigned to postconditioning arm (primary angioplasty (PA) and stenting followed by brief episodes of ischemia-reperfusion performed during the first minutes of reperfusion) or non-postconditioning arm (PA and stenting without additional intervention). All patients will be treated medically according to current international guidelines, including glycoprotein IIb/IIIa inhibitors before PCI. The primary end point is to evaluate whether postconditioning, compared to PA without additional intervention, reduces infarct size estimated by magnetic resonance at 30±10 days after the AMI. Secondary end points are microvascular obstruction observed at magnetic resonance, ST-segment elevation resolution, persistent ST-segment elevation, angiographic myocardial blush grade <2 and non sustained/sustained ventricular tachycardia in the 48 hours following PA. Further secondary end points are enzymatic infarct size, left ventricular remodeling and left ventricular function at magnetic resonance performed at 6±1 months, and the reduction of major adverse cardiac events at 30 days and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* clinical evidence of myocardial infarction defined by the presence of ischemic chest pain lasting more than 30 minutes, with a time interval from the onset of symptoms less than 6 hours before hospital admission, associated with typical ST-segment elevation on the 12-lead ECG
* angiographic-detected culprit lesion with stenosis diameter >70% and TIMI flow grade <=1

Exclusion Criteria:

* previous acute myocardial infarction
* previous myocardial revascularization (angioplasty or coronary bypass)
* previous heart valve replacement
* previous heart transplant
* clinical instability precluding the suitability of the study
* cardiogenic shock or persistent hypotension (systolic blood pressure <100 mmHg)
* rescue angioplasty after thrombolytic therapy
* evidence of coronary collaterals (Rentrop grade>0) in the risk area
* advanced atrioventricular block
* significant bradycardia
* absence of sinus rhythm
* inability to lay flat (due to severe cardiac heart failure/respiratory insufficiency)
* history or clinical evidence of bronchospastic lung disease
* pregnancy
* known existence of a life-threatening disease with a life expectancy <6 months
* inability to give informed consent
* any contraindication to undergo cardiac-MRI, such as implanted metallic objects (cardiac pacemakers and/or implantable cardioverter defibrillator, implanted insulin pumps or any other type of electronic devices, cerebral clips, aneurysm clips) or any other contraindication to cardiac-MRI (such as claustrophobia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2007-04; Primary Completion 2010-01 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Infarct size estimated by magnetic resonance | 30±10 days after myocardial infartion

SECONDARY OUTCOMES:
Microvascular obstruction observed at magnetic resonance | 30±10 days after myocardial infarction
ST-segment elevation resolution | First post-intervention ECG
Persistent ST-segment elevation | At 24 and 48 hours post-intervention ECG
Angiographic myocardial blush grade <2 | After primary angioplasty
Non sustained/sustained ventricular tachycardia | Within 48 hours after miocardial infarction
Enzymatic infarct size | Within 7 days after myocardial infarction
Left ventricular remodeling and left ventricular function at MRI | At 6±1 months
Incidence of Major Adverse Cardiac Events (MACE), defined as the combination of death, re-infarction, re-hospitalization for heart failure or repeat revascularization | At 30 days and at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Tarantini, MD, Ph.D., Principal Investigator — Department of Cardiac, Thoracic and Vascular Sciences, University of Padua
Locations (1):
- Department of Cardiac, Thoracic and Vascular Sciences, University of Padua, Italy, Padua, Italy

REFERENCES:
- [Background] Thom T, Haase N, Rosamond W, Howard VJ, Rumsfeld J, Manolio T, Zheng ZJ, Flegal K, O'Donnell C, Kittner S, Lloyd-Jones D, Goff DC Jr, Hong Y, Adams R, Friday G, Furie K, Gorelick P, Kissela B, Marler J, Meigs J, Roger V, Sidney S, Sorlie P, Steinberger J, Wasserthiel-Smoller S, Wilson M, Wolf P; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2006 update: a report from the American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Circulation. 2006 Feb 14;113(6):e85-151. doi: 10.1161/CIRCULATIONAHA.105.171600. Epub 2006 Jan 11. No abstract available. PMID 16407573
- [Background] Reffelmann T, Hale SL, Li G, Kloner RA. Relationship between no reflow and infarct size as influenced by the duration of ischemia and reperfusion. Am J Physiol Heart Circ Physiol. 2002 Feb;282(2):H766-72. doi: 10.1152/ajpheart.00767.2001. PMID 11788428
- [Background] Vinten-Johansen J, Yellon DM, Opie LH. Postconditioning: a simple, clinically applicable procedure to improve revascularization in acute myocardial infarction. Circulation. 2005 Oct 4;112(14):2085-8. doi: 10.1161/CIRCULATIONAHA.105.569798. No abstract available. PMID 16203924
- [Background] Staat P, Rioufol G, Piot C, Cottin Y, Cung TT, L'Huillier I, Aupetit JF, Bonnefoy E, Finet G, Andre-Fouet X, Ovize M. Postconditioning the human heart. Circulation. 2005 Oct 4;112(14):2143-8. doi: 10.1161/CIRCULATIONAHA.105.558122. Epub 2005 Sep 26. PMID 16186417
- [Background] Ottani F, Galvani M, Ferrini D, Sorbello F, Limonetti P, Pantoli D, Rusticali F. Prodromal angina limits infarct size. A role for ischemic preconditioning. Circulation. 1995 Jan 15;91(2):291-7. doi: 10.1161/01.cir.91.2.291. PMID 7805230
- [Background] Kloner RA, Shook T, Antman EM, Cannon CP, Przyklenk K, Yoo K, McCabe CH, Braunwald E. Prospective temporal analysis of the onset of preinfarction angina versus outcome: an ancillary study in TIMI-9B. Circulation. 1998 Mar 24;97(11):1042-5. doi: 10.1161/01.cir.97.11.1042. PMID 9531250
- [Background] Smith SC Jr, Feldman TE, Hirshfeld JW Jr, Jacobs AK, Kern MJ, King SB 3rd, Morrison DA, O'Neill WW, Schaff HV, Whitlow PL, Williams DO, Antman EM, Adams CD, Anderson JL, Faxon DP, Fuster V, Halperin JL, Hiratzka LF, Hunt SA, Nishimura R, Ornato JP, Page RL, Riegel B; American College of Cardiology/American Heart Association Task Force on Practice Guidelines; American College of Cardiology/American Heart Association/Society for Cardiovascular Angiography and Interventions Writting Committee to Update the 2001 Guidelines for Percutaneous Coronary Intervention. ACC/AHA/SCAI 2005 Guideline Update for Percutaneous Coronary Intervention--summary article: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines (ACC/AHA/SCAI Writing Committee to Update the 2001 Guidelines for Percutaneous Coronary Intervention). Circulation. 2006 Jan 3;113(1):156-75. doi: 10.1161/CIRCULATIONAHA.105.170815. No abstract available. PMID 16391169
- [Background] van 't Hof AW, Liem A, Suryapranata H, Hoorntje JC, de Boer MJ, Zijlstra F. Angiographic assessment of myocardial reperfusion in patients treated with primary angioplasty for acute myocardial infarction: myocardial blush grade. Zwolle Myocardial Infarction Study Group. Circulation. 1998 Jun 16;97(23):2302-6. doi: 10.1161/01.cir.97.23.2302. PMID 9639373
- [Background] Svilaas T, van der Horst IC, Zijlstra F. Thrombus Aspiration during Percutaneous coronary intervention in Acute myocardial infarction Study (TAPAS)--study design. Am Heart J. 2006 Mar;151(3):597.e1-597.e7. doi: 10.1016/j.ahj.2005.11.010. PMID 16504620
- [Background] Kim RJ, Shah DJ, Judd RM. How we perform delayed enhancement imaging. J Cardiovasc Magn Reson. 2003 Jul;5(3):505-14. doi: 10.1081/jcmr-120022267. PMID 12882082
- [Background] Cerqueira MD, Weissman NJ, Dilsizian V, Jacobs AK, Kaul S, Laskey WK, Pennell DJ, Rumberger JA, Ryan T, Verani MS; American Heart Association Writing Group on Myocardial Segmentation and Registration for Cardiac Imaging. Standardized myocardial segmentation and nomenclature for tomographic imaging of the heart. A statement for healthcare professionals from the Cardiac Imaging Committee of the Council on Clinical Cardiology of the American Heart Association. Circulation. 2002 Jan 29;105(4):539-42. doi: 10.1161/hc0402.102975. No abstract available. PMID 11815441
- [Background] Judd RM, Lugo-Olivieri CH, Arai M, Kondo T, Croisille P, Lima JA, Mohan V, Becker LC, Zerhouni EA. Physiological basis of myocardial contrast enhancement in fast magnetic resonance images of 2-day-old reperfused canine infarcts. Circulation. 1995 Oct 1;92(7):1902-10. doi: 10.1161/01.cir.92.7.1902. PMID 7671375
- [Background] Lima JA, Judd RM, Bazille A, Schulman SP, Atalar E, Zerhouni EA. Regional heterogeneity of human myocardial infarcts demonstrated by contrast-enhanced MRI. Potential mechanisms. Circulation. 1995 Sep 1;92(5):1117-25. doi: 10.1161/01.cir.92.5.1117. PMID 7648655
- [Background] Braunwald E, Domanski MJ, Fowler SE, Geller NL, Gersh BJ, Hsia J, Pfeffer MA, Rice MM, Rosenberg YD, Rouleau JL; PEACE Trial Investigators. Angiotensin-converting-enzyme inhibition in stable coronary artery disease. N Engl J Med. 2004 Nov 11;351(20):2058-68. doi: 10.1056/NEJMoa042739. Epub 2004 Nov 7. PMID 15531767
- [Derived] Tarantini G, Favaretto E, Marra MP, Frigo AC, Napodano M, Cacciavillani L, Giovagnoni A, Renda P, De Biasio V, Plebani M, Mion M, Zaninotto M, Isabella G, Bilato C, Iliceto S. Postconditioning during coronary angioplasty in acute myocardial infarction: the POST-AMI trial. Int J Cardiol. 2012 Dec 15;162(1):33-8. doi: 10.1016/j.ijcard.2012.03.136. Epub 2012 Apr 9. PMID 22494866
- [Derived] Tarantini G, Favaretto E, Napodano M, Perazzolo Marra M, Cacciavillani L, Babuin L, Giovagnoni A, Renda P, De Biasio V, Plebani M, Mion M, Zaninotto M, Mistrorigo F, Panfili M, Isabella G, Bilato C, Iliceto S. Design and methodologies of the POSTconditioning during coronary angioplasty in acute myocardial infarction (POST-AMI) trial. Cardiology. 2010;116(2):110-6. doi: 10.1159/000316967. Epub 2010 Jun 29. PMID 20588019